CLINICAL TRIAL: NCT06758388
Title: The Relationship Between Physical and Psychosocial Status and Irisin Level in Individuals With Knee Osteoarthritis Performing Brisk Walking Exercise
Brief Title: Exercise-induced Irisin in Individuals With Knee Osteoarthritis.
Acronym: Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ümmahani Kuş (Other)
Responsible Party: Sponsor-Investigator, Ümmahani Kuş, Investigator, Alanya Alaaddin Keykubat University
Organization: Alanya Alaaddin Keykubat University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-11095095-050.04-225853
Record Dates: First submitted 2024-12-12; First posted 2025-01-03 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis (Knee OA)
Keywords: Knee osteoarthritis; İrisin; FNDC5; Pain; Functional capacity; Depression; Fatigue; Sleep quality; Quality of life; Muscle strength
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Depression; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Other): The control group will perform a home exercise program that includes progressive strengthening exercises.
  Interventions: Other: home exercise program
- Intervention group (Active Comparator): The intervention group will perform a home exercise program that includes progressive strengthening exercises and brisk walking exercise.
  Interventions: Behavioral: home exercise program + brisk walking exercise

INTERVENTIONS:
Other: home exercise program — The prepared home exercise program is a program that includes gradual strengthening exercises that participants will do once a day, 5 days a week, for 8 weeks. The exercises will be performed as 1 set for the first 2 weeks, 2 sets in the 3rd and 4th weeks, and 3 sets in the last 4 weeks.
  Arms: Control group
Behavioral: home exercise program + brisk walking exercise — In addition to the home exercise program applied by the control group, a brisk walk will be performed. The brisk walking exercise will be done for 30 minutes, 5 days a week for 8 weeks. The intensity of the exercise will be adjusted according to the Borg CR-10 scale and the Speech test. Moderate intensity exercise is recommended for participants. The participant will walk rhythmically for 30 minutes at a speed where he/she will give 4-6 points on the Borg CR-10 Scale, and can speak a few sentences without getting out of breath according to the Speech test, but cannot sing. Before and after the brisk walk, he/she will be asked to walk at a slow speed for 5 minutes (warm-up-cool down).
  Arms: Intervention group

SUMMARY:
The goal of this prospective randomised controled study is to investigate the effect of 8-weeks brisk walking exercise on irisin levels, physical and psychosocial parameters in individuals with knee osteoarthritis, and the relationship between irisin levels and physical and psychosocial parameters. The main question it aims to answer is: does 8-weeks brisk walking exercise increase irisin levels and imoroves physical and psychosocial parameters and is the irisin level in relation with the physical and psychosocial parameters.

DETAILED DESCRIPTION:
Irisin is a myokine secreted by skeletal muscle after physical activity. It improves subchondral bone density and quality by increasing osteoblast differentiation and proliferation and improves the mechanical support of cartilage. In addition, irisin promotes chondrocyte proliferation, inhibits chondrocyte apoptosis, and reduces the secretion of inflammatory factors and matrix metalloproteinases. As a result of all these, improvements in joint function may be achieved.

Besides, irisin can improve depressive mood in patients with depression, and irisin level is found to be positively correlated with sleep quality and negatively correlated with disease duration and disease activity in patients with rheumatoid arthritis.

This study aims to investigate the effect of an 8-week moderate-intensity brisk walking exercise program on irisin serum levels and physical and psychosocial parameters in individuals with knee osteoarthritis and the relationship between irisin levels and physical and psychosocial parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic knee OA
* Stage 1-3 knee OA according to the Kellgren-Lawrence classification
* Patients aged 40-65
* Patients agreeing to participate in the study
* Patients having physical and cognitive ability to participate in the exercise program

Exclusion Criteria:

* History of depression and/or anxiety etc. psychiatric disease
* Uncontrolled hypertension, uncontrolled heart rhythm disorders, history of hospitalization for cardiovascular reasons in the last 6 months
* History of symptomatic pulmonary disease
* Use of medication due to dyslipidemia and/or diabetes
* Presence of acute inflammation or effusion in the knee joint
* Presence of central or peripheral neurological disease that will cause loss of lower extremity muscle strength, sensation, and balance
* Presence of a prosthetic joint in the knee and previous lower extremity surgery
* Having received a physical therapy program in the last 6 months
* Patients with severe visual or hearing impairment
* Patients with severe peripheral vascular disorders
* Presence of severe knee joint instability, ligament and meniscal damage
* Being illiterate

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 8 weeks
  The most commonly used measurement tool to assess pain is the Visual Analog Scale (VAS). Patients are asked to rate the intensity of their pain at rest and during activity. A score of 0 indicates no pain, while a score of 10 indicates unbearable pain.
Range of Motion of the Joint | 8 weeks
  To measure the range of motion of knee flexion and extension, the pivot point of the goniometer is the lateral condyle of the femur while the patient is in the prone position. One of the arms of the goniometer is fixed parallel to the lateral midline of the femur. The movable arm follows the fibula. The degree that the patient can perform is recorded.
Muscle Strength | 8 weeks
  Quadriceps muscle strength will be assessed with a hand-held dynamometer (Lafayette). The participant is in a sitting position with hips and knees flexed to 90°. The dynamometer is placed on the anterior surface of the leg just proximal to the ankle. During the measurement, the participant is asked to apply maximum pushing force against the device for 5 seconds. The measured force will be recorded in 'kg'.
Functional Level | 8 weeks
  The six-minute walk test (6MWT) will be used to determine the functional level. The 6MWT is used to evaluate the person's endurance and ability to walk long distances. The person walks the maximum distance they can walk as fast as possible on a 30-meter flat track in 6 minutes. The distance the person walked is added up at the end of the test and the longer distance indicates better performance.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 8 weeks
  KOOS is a self-report scale used to assess symptoms and functional status that may develop due to knee injuries and osteoarthritis. The scale, which questions the last week, has 5 subgroups: symptoms, pain, functional status related to daily living activities, functional status in sports and leisure activities, and quality of life related to the knee, and the scale consists of a total of 42 questions. Each subsection is scored between 0 and 100 points, with 0 points indicating a serious problem and 100 points indicating no problem.
Assessment of quality of life | 8 weeks
  The Knee and Hip Osteoarthritis Quality of Life Scale (OAKHQOL) will be used to assess quality of life. The Knee and Hip Osteoarthritis Quality of Life Scale consists of 5 subsections: physical activity, mental health, pain, social functions and social support. The scale consists of 43 items. Each item in the scale is scored between 0 and 10, taking into account the last 4 weeks. 0 means 'not at all', 10 means 'very extreme, constant'. The calculation is made out of 100 according to the average score of the items in each subsection. As the total score increases, the quality of life increases.
Depression | 8 weeks
  The presence of depression will be assessed with the Beck Depression Index-II (BDI-II). The BDI-II consists of 21 items. Participants are asked to give a score between 0 and 3 for each item, taking into account the last week. The severity of depression increases as the total score obtained from the scale increases. The main difference between the BDI-II and previous versions is that it includes items that aim to measure structures such as loss of energy, worthlessness, appetite disorders and concentration.
Fatigue | 8 weeks
  The Fatigue Severity Scale will be used to assess fatigue. The Fatigue Severity Scale assesses fatigue in the last month. The scale consists of 9 items and the items are scored between 0 and 7. A score of 0 means I completely disagree, a score of 7 means I agree. The scale score is obtained by dividing the total score by the number of items. The higher the score, the higher the fatigue level.
Sleep Quality | 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI) will be used to assess sleep quality. The scale, which assesses the person's sleep quality in the last month, begins with 4 open-ended questions and consists of a total of 24 questions. In the PSQI assessment, 18 questions answered by the person themselves are used in scoring. The PSQI has 7 components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, sleeping pill use, and daytime dysfunction. Each question is answered on a scale of 0-3. The sum of the 7 component scores constitutes the total PSQI score. The total score of the scale is between 0 and 21 points. A total score of 5 or less indicates good sleep quality, while a score above 5 indicates poor sleep quality.
İrisin level | 8 weeks
  Blood samples will be collected from the participants at the beginning of the study and after 8 weeks of exercise (1 day after the last exercise). Blood samples will be centrifuged at 3000 rpm at +4 0C for 10 minutes to separate plasma and samples will be collected in aliquots in Eppendorf tubes and stored at -80 0C until the day of the study. Serum irisin level will be determined using the human irisin Enzyme-Linked Immunosorbent Assay (ELISA) test kit.
Body mass index | 8 weeks
  Weight and height will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
Correlation between irisin level (ng/mL) and primary outcome measures | 8 weeks
  Multivariate analyses will be carried out with control variables;
  * Body mass index (Weight and height will be combined to report BMI in kg/m^2)
  * Pain VAS score
  * Quadriceps strength assessed with hand-held dynamometer (HHD) (Kg)
  * Six-minute walk test (m)
  * Knee Injury and Osteoarthritis Outcome Score
  * The Knee and Hip Osteoarthritis Quality of Life Scale (OAKHQOL) Score
  * Beck Depression Index-II (BDI-II) Score
  * Fatigue Severity Scale Score
  * Pittsburgh Sleep Quality Index (PSQI) Score
  * Range of motion (degrees)

CONTACTS AND LOCATIONS:
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes